CLINICAL TRIAL: NCT01075906
Title: An Open-label, Parallel-group, Multiple-Dose, Pharmacokinetic and Safety Study of Colchicine Pediatric Formulation in Pediatric and Adult Patients With FMF
Brief Title: Pharmacokinetics Study of Colchicine in Familial Mediterranean Fever (FMF) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-006-09-1001
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Familial Mediterranean Fever
Keywords: pharmacokinetics
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine Sprinkle Capsules, 0.3 mg - dose administered according to age range on Day 1
  Interventions: Drug: colchicine sprinkle capsules
- colchicine at steady state (Experimental): colchicine sprinkle capsules 0.3 mg - dose administered according to age range on Day 15 following once daily dosing of colchicine on Days 2 - 14
  Interventions: Drug: colchicine sprinkle capsules

INTERVENTIONS:
Drug: colchicine sprinkle capsules — 0.3 mg
  Arms: Colchicine
Drug: colchicine sprinkle capsules — 0.3 mg
  Arms: colchicine at steady state

SUMMARY:
Colchicine is widely recognized as safe and effective treatment of Familial Mediterranean Fever (FMF) in children and adults. Colchicine is currently used to treat FMF in younger patients by inexact dosing through breaking or crushing adult-dose tablets. An age-appropriate sprinkle formulation will allow for more accurate dosing in pediatric patients. The primary objective of this study is to evaluate and compare the steady-state pharmacokinetics of multiple oral doses of colchicine sprinkle capsules administered to pediatric and adult FMF patients.

Secondary objectives include evaluation of the safety and tolerability of this regimen in pediatric and adult FMF patients and measurement of the levels of acute phase reactants (i.e, serum amyloid A [SAA], erythrocyte sedimentation rate [ESR], C-reactive protein [CRP]) at baseline and after dosing.

DETAILED DESCRIPTION:
FMF patients who have not been taking colchicine (colchicine-naïve patients) will be enrolled into a 1 week dose-titration period (Days -7 to -1). Beginning on Day -7, a pre-dose blood sample will be collected from the colchicine-naïve patient population for determination of pharmacodynamic markers. Patients will then be administered a low starting dose of colchicine (as determined by the principal investigator) titrated up to the study colchicine dose which is 0.6 mg (2 capsules) in children ≥2 to < 6 years old, 0.9 mg (3 capsules) in children ≥6 to < 12, 1.2 mg (4 capsules) in children ≥12 to < 16 and adults ≥16 and < 65. On Day 2, patients will return to the clinic for collection of a pre-dose blood sample followed by administration of the study dose of colchicine. On Days 3-7, patients (parent/guardian) will self-medicate with the study dose of colchicine recording the time of dosing and any adverse events. On Days 8-14, patients (parent/guardian) will self-medicate with the study dose of colchicine recording the time of dosing and any adverse events. On the morning of Day 15, patients will return to the clinic for collection of a pre-dose blood sample followed by administration of the study dose of colchicine. Blood samples will be collected post-dose at times sufficient to adequately define the pharmacokinetics of colchicine and its metabolites. Safety and tolerability of this dosing regimen will be determined by evaluation of vital signs and adverse events during the study and upon completion of the study. All adverse events will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 2-65 years with a confirmed clinical diagnosis of FMF,
* Non-pregnant, and
* If of child-bearing potential, using effective contraceptive measures.

Exclusion Criteria:

* Recent participation (within 30 days) in other research studies,
* Pregnant or lactating,
* History or current infection of human immunodeficiency virus (HIV), hepatitis A, B or C,
* Current or recent use of any drugs/drug classes or combinations thereof that may affect the absorption or metabolism of colchicine,
* Clinically relevant abnormal clinical laboratories at screening,
* Current or recent (<6 months) history of severe, unstable or uncontrolled neurological, cardiovascular, gastrointestinal, hematological, moderate or severe hepatic and/or renal disease, or evidence of other diseases at the physical examination conducted at the screening.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration | 15 days
  pharmacokinetic samples collected pre-dose on Days 1, 2 and 15 and at 0.25 - 0.5 hours, 1.5-2.5 hours and at 5-8 hours post-dose on Days 1 and 15
Area Under the Concentration Time Curve from Time Zero to the Time of Last Measured Concentration (AUC 0-t) | 15 days
  Pharmacokinetic samples collected pre-dose on Days 1,2 and 15 and at 0.25-0.5 hours, 1.5-2.5 hours and 5-8 hours post-dose on Days 1 and 15.
Area Under the Concentration Time Curve from Zero through Infinity | 15 days
  Pharmacokinetic samples collected pre-dose on Days 1, 2 and 15 and at 0.25-0.5 hours, 1.5-2.5 hours and at 5-8 hours post-dose on Days 1 and 15

SECONDARY OUTCOMES:
Acute Phase Reactant (ESR, CRP, SAA) Levels | 15 days
  Pharmacodynamic samples collected pre-dose on Days 7, 1 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davis, MD, Study Chair — Mutual Pharmaceutical Company, Inc.
Locations (10):
- Childrens Hospital Los Angeles, Los Angeles, California, United States
- Center of Medical Genetics and Primary Health Care, Yerevan, Yerevan, Armenia
- Israel (6):
  - Soroka Medical Center, Beersheba, Beer Sheba
  - Rambam Medical Center, Haifa, Haifa District
  - Hadassah Medical Center, Jerusalem, Israel
  - Pediatric Rheumatology Unit - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Safra Children's Hospital, Tel Litwinsky, Tel Hashomer
  - Sheba Medical Center, Tel Litwinsky, Tel Hashomer
- Turkey (Türkiye) (2):
  - Hacettepe University, Ankara, Ankara
  - Cerrahpasa Medical Facility, Istanbul, Istanbul